CLINICAL TRIAL: NCT02825251
Title: Efficacy and Safety of Continuous Subcutaneous Insulin Infusion of Faster-acting Insulin Aspart Compared to NovoRapid® in Adults With Type 1 Diabetes
Acronym: Onset® 5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN1218-3854; 2010-024054-11 (EudraCT Number); U1111-1118-2480 (Other: WHO); NL54555.018.16 (Other: CCMO)
Record Dates: First submitted 2016-07-04; First posted 2016-07-07 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Faster-acting insulin aspart CSII (Experimental)
  Interventions: Drug: Faster-acting insulin aspart
- NovoRapid® CSII (Active Comparator)
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: Faster-acting insulin aspart — Injected s.c. /subcutaneously (under the skin)
  Arms: Faster-acting insulin aspart CSII
Drug: insulin aspart — Injected s.c. /subcutaneously (under the skin)
  Arms: NovoRapid® CSII

SUMMARY:
This trial is conducted in Europe and the United States of America (USA). The aim of this trial is to investigate efficacy and safety of Continuous Subcutaneous Insulin Infusion of Faster-acting Insulin Aspart compared to NovoRapid® in Adults with Type 1 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age at least 18 years at the time of signing the informed consent
* Diagnosed with T1DM (Type 1 Diabetes Mellitus) (based on clinical judgement and/or supported by laboratory analysis as per local guidelines) equal or above 1 year prior to the day of screening
* Using the same Medtronic pump (Minimed 530G (551/751), Paradigm Veo (554/754), Paradigm Revel (523/723), Paradigm (522/722)) for CSII in a basal-bolus regimen with a rapid acting insulin analogue for at least six months prior to screening and willing to stay on the same pump model throughout the trial (if the model is changed the change should not exceed 7 consecutive days.)
* HbA1c (glycosylated haemoglobin) 7.0-9.0% (53-75 mmol/mol) as assessed by central laboratory at screening
* Body mass index (BMI) below or equal to 35.0 kg/m^2 at screening
* Ability and willingness to take at least 3 daily meal-time insulin bolus infusions every day throughout the trial

Exclusion Criteria:

* Any of the following: myocardial infarction, stroke, hospitalization for unstable angina or transient ischaemic attack within the past 180 days prior to the day of screening
* Planned coronary, carotid or peripheral artery revascularisation known on the day of screening
* History of hospitalization for ketoacidosis below or equal to 180 days prior to the day of screening
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria in a period of 90 days before screening
* Any condition which, in the opinion of the Investigator, might jeopardise a Subject's safety or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2016-07-06 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (86):
- United States (28):
  - Novo Nordisk Investigational Site, Encino, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Roseville, California
  - Novo Nordisk Investigational Site, San Mateo, California
  - Novo Nordisk Investigational Site, San Ramon, California
  - Novo Nordisk Investigational Site, Santa Barbara, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Newark, Delaware
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Idaho Falls, Idaho
  - Novo Nordisk Investigational Site, Arlington Heights, Illinois
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Asheville, North Carolina
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Amarillo, Texas
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Mesquite, Texas
  - Novo Nordisk Investigational Site, Federal Way, Washington
  - Novo Nordisk Investigational Site, Renton, Washington
- Belgium (7):
  - Novo Nordisk Investigational Site, Arlon
  - Novo Nordisk Investigational Site, Bonheiden
  - Novo Nordisk Investigational Site, Brussels
  - Novo Nordisk Investigational Site, Edegem
  - Novo Nordisk Investigational Site, Leuven
  - Novo Nordisk Investigational Site, Sint-Niklaas
  - Novo Nordisk Investigational Site, Wilrijk
- Canada (8):
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Barrie, Ontario
  - Novo Nordisk Investigational Site, Concord, Ontario
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Oakville, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Montreal, Quebec
  - Novo Nordisk Investigational Site, Québec
- France (10):
  - Novo Nordisk Investigational Site, Caen
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Le Creusot
  - Novo Nordisk Investigational Site, Montpellier
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Saint-Herblain
  - Novo Nordisk Investigational Site, Strasbourg
  - Novo Nordisk Investigational Site, Toulouse
  - Novo Nordisk Investigational Site, Vénissieux
- Germany (9):
  - Novo Nordisk Investigational Site, Bad Mergentheim
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Friedrichsthal
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Ludwigshafen
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Neuwied
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Rostock
- Netherlands (10):
  - Novo Nordisk Investigational Site, Amsterdam
  - Novo Nordisk Investigational Site, Apeldoorn
  - Novo Nordisk Investigational Site, Eindhoven
  - Novo Nordisk Investigational Site, Hoofddorp
  - Novo Nordisk Investigational Site, Hoogeveen
  - Novo Nordisk Investigational Site, Leiden
  - Novo Nordisk Investigational Site, Nijmegen
  - Novo Nordisk Investigational Site, Rotterdam
  - Novo Nordisk Investigational Site, Utrecht
  - Novo Nordisk Investigational Site, Venlo
- Russia (6):
  - Novo Nordisk Investigational Site, Cheboksary
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Saratov
  - Novo Nordisk Investigational Site, Yoshkar-Ola
- Slovenia (2):
  - Novo Nordisk Investigational Site, Ljubljana
  - Novo Nordisk Investigational Site, Novo Mesto
- United Kingdom (6):
  - Novo Nordisk Investigational Site, Cambridge
  - Novo Nordisk Investigational Site, Guildford
  - Novo Nordisk Investigational Site, Harrogate, North Yorkshire
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Manchester
  - Novo Nordisk Investigational Site, St Helens

REFERENCES:
- [Result] Zijlstra E, Demissie M, Graungaard T, Heise T, Nosek L, Bode B. Investigation of Pump Compatibility of Fast-Acting Insulin Aspart in Subjects With Type 1 Diabetes. J Diabetes Sci Technol. 2018 Jan;12(1):145-151. doi: 10.1177/1932296817730375. Epub 2017 Sep 18. PMID 28918652
- [Result] Klonoff DC, Evans ML, Lane W, Kempe HP, Renard E, DeVries JH, Graungaard T, Hyseni A, Gondolf T, Battelino T. A randomized, multicentre trial evaluating the efficacy and safety of fast-acting insulin aspart in continuous subcutaneous insulin infusion in adults with type 1 diabetes (onset 5). Diabetes Obes Metab. 2019 Apr;21(4):961-967. doi: 10.1111/dom.13610. Epub 2019 Jan 13. PMID 30537180
- [Derived] Gorst-Rasmussen A, Sturis J, Ekelund M. Continuous Glucose Monitoring Sensor Glucose Levels and Insulin Pump Infusion Set Wear-Time During Treatment with Fast-Acting Insulin Aspart: A Post Hoc Analysis of Onset 5. Diabetes Technol Ther. 2022 Jan;24(1):10-17. doi: 10.1089/dia.2021.0199. Epub 2021 Dec 14. PMID 34524005
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 92 sites in 9 countries.as follows: Belgium (7), Canada (8), France (10), Germany (9), Netherlands (9), Russian Federation (11), Slovenia (2), United Kingdom (6), and United States (30). One (1) site in the Netherlands screened, but didn't randomise any subject.
Pre-assignment Details: There was a 4-week run-in period primarily for reinforcement of subject training in trial procedures, diabetes education and collecting baseline assessments. Subjects remained on their pre-trial insulin treatment during the run-in period.
Groups:
- Faster Aspart: The subjects received faster aspart (basal-bolus regimen) by continuous subcutaneous insulin infusion (CSII) for 16 weeks. Doses of basal and bolus insulin and timing of bolus dose were individually adjusted and thus no maximum dose of insulin was specified. Basal rate insulin adjustment: The purpose of adjusting the basal rates was to ensure that blood glucose (BG) was kept between 4.0-6.0 mmol/L [71-108 mg/dL] while in a fasting state and during the night. Bolus insulin titration: It was recommended that meal-time bolus insulin was titrated based on carbohydrate-counting using the Bolus Wizard® according to their usual practice and according to instructions from the investigator. Meal-time dosing was defined as bolus infusion initiated 0-2 minutes before a meal.
- NovoRapid: The subjects received insulin aspart (NovoRapid®/NovoLog®: basal-bolus regimen) by CSII for 16 weeks. Doses of basal and bolus insulin and timing of bolus dose were individually adjusted and thus no maximum dose of insulin was specified. Basal rate insulin adjustment: The purpose of adjusting the basal rates was to ensure that BG was kept between 4.0-6.0 mmol/L [71-108 mg/dL] while in a fasting state and during the night. Bolus insulin titration: It was recommended that meal-time bolus insulin was titrated based on carbohydrate-counting using the Bolus Wizard® according to their usual practice and according to instructions from the investigator. Meal-time dosing was defined as bolus infusion initiated 0-2 minutes before a meal.
Period: Overall Study
Arm/Group | Faster Aspart | NovoRapid
Started | 236 | 236
Completed | 233 | 230
Not Completed | 3 | 6
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Unclassified | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Faster Aspart: The subjects received faster aspart (basal-bolus regimen) by CSII for 16 weeks. Doses of basal and bolus insulin and timing of bolus dose were individually adjusted and thus no maximum dose of insulin was specified. Basal rate insulin adjustment: The purpose of adjusting the basal rates was to ensure that BG was kept between 4.0-6.0 mmol/L [71-108 mg/dL] while in a fasting state and during the night. Bolus insulin titration: It was recommended that meal-time bolus insulin was titrated based on carbohydrate-counting using the Bolus Wizard® according to their usual practice and according to instructions from the investigator. Meal-time dosing was defined as bolus infusion initiated 0-2 minutes before a meal.
- Total: Total of all reporting groups
Arm/Group | Faster Aspart | NovoRapid | Total
Number analyzed (Participants) | 236 | 236 | 472
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The full analysis (FAS) included all randomised subjects.
  Years | 43.3 (14.8) | 43.6 (14.7) | 43.5 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The FAS included all randomised subjects.
  Participants
    Female | 133 | 136 | 269
    Male | 103 | 100 | 203
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The FAS included all randomised subjects.
  Participants
    Hispanic or Latino | 7 | 6 | 13
    Not Hispanic or Latino | 210 | 215 | 425
    Unknown or Not Reported | 19 | 15 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The FAS included all randomised subjects.
  Participants
    American Indian or Alaska Native | 0 | 2 | 2
    Asian | 3 | 3 | 6
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 5 | 7
    White | 209 | 210 | 419
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 22 | 16 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change from baseline (week 0) in HbA1c was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period. In-trial period: the observation period from date of randomisation until last trial-related subject-site contact.
Time Frame: Week 0, week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: Percentage (%) of HbA1c
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Percentage (%) of HbA1c
  Baseline | 7.49 (0.55) | 7.49 (0.53)
  Change from baseline | -0.06 (0.50) | -0.14 (0.44)
Statistical Analysis 1: Comparison: Faster Aspart vs NovoRapid; Change from baseline in HbA1c was analysed using an analysis of variance model after multiple imputation assuming treatment according to randomisation. The model included treatment, strata (use of own continuous glucose monitoring), previous insulin use, and region as factors, and baseline HbA1c as a covariate; Test type: Non-Inferiority — Non-inferiority of faster aspart was considered confirmed if the upper limit of the two-sided 95 % CI for the true treatment-difference D (faster aspart minus NovoRapid®) was below 0.4 %; ANOVA; Treatment difference = 0.09, 95% CI 2-sided [0.01 to 0.17]

2. Secondary Outcome: Change From Baseline in 1-hour PPG Increment
Description: Change from baseline (week 0) in 1-hour postprandial glucose (PPG) increment was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, Week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L
  Baseline: number analyzed (Participants) | 235 | 235
  Baseline | 4.67 (3.09) | 4.62 (3.00)
  Change from baseline: number analyzed (Participants) | 228 | 227
  Change from baseline | -0.89 (3.44) | 0.05 (3.37)

3. Secondary Outcome: Change From Baseline in 1,5-anhydroglucitol
Description: Change from baseline (week 0) in 1,5-anhydroglucitol was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, Week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
ug/mL
  Baseline: number analyzed (Participants) | 233 | 234
  Baseline | 4.20 (2.34) | 4.13 (2.14)
  Change from baseline: number analyzed (Participants) | 233 | 234
  Change from baseline | 0.14 (1.48) | 0.25 (1.42)

4. Secondary Outcome: Change From Baseline in Time Spent in Low IG (≤3.9 mmol/L [70 mg/dL]) During CGM
Description: Change from baseline (week 0) in low interstitial glucose (IG) (≤3.9 mmol/L [70 mg/dL]) during continuous glucose monitoring (CGM) was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: min/day
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
min/day
  Baseline | 85.42 (65.20) | 79.88 (60.46)
  Change from baseline: number analyzed (Participants) | 234 | 231
  Change from baseline | -6.96 (55.29) | 2.85 (58.56)

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Change from baseline (week 0) in FPG was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L
  Baseline: number analyzed (Participants) | 231 | 233
  Baseline | 7.60 (2.64) | 7.40 (2.31)
  Change from baseline: number analyzed (Participants) | 231 | 233
  Change from baseline | -0.03 (3.19) | 0.25 (3.05)

6. Secondary Outcome: Percentage of Subjects Reaching HbA1c <7.0% (53 mmol/Mol)
Description: Percentage of subjects reaching HbA1c <7.0% (53 mmol/mol) was evaluated after 16 weeks of randomisation. Subjects without an HbA1c measurement at week 16 were considered not to have achieved HbA1c target at week 16. The results are based on the in-trial period.
Time Frame: Week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Number; unit: % of subjects
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
% of subjects | 20.3 | 23.3

7. Secondary Outcome: Percentage of Subjects Reaching HbA1c <7.0% (53 mmol/Mol) Without Severe Hypoglycaemic Episodes
Description: Percentage of subjects reaching HbA1c <7.0% (53 mmol/mol) without treatment emergent severe hypoglycaemic episodes was evaluated after 16 weeks of randomisation. Subjects without an HbA1c measurement at week 16 were considered not to have achieved HbA1c target at week 16. Severe hypoglycaemia: An episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. Plasma glucose (PG) concentrations may not be available during an event, but neurological recovery following the return of PG to normal was considered sufficient evidence that the event was induced by a low PG concentration. Treatment emergent: hypoglycaemic episodes were defined as treatment emergent if the onset of the episode occurred on or after the first day of IMP administration after randomisation (in week 0) and no later than one day after the last day on IMP (i.e., maximum week 16 + 1 day). The results are based on the in-trial period.
Time Frame: Week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Number; unit: % of subjects
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
% of subjects | 18.6 | 22.5

8. Secondary Outcome: Change From Baseline in 30-min, 1-hour, 2-hour, 3-hour and 4-hour PPG (Meal Test)
Description: Change from baseline (week 0) in 30-minute, 1-hour, 2-hour, 3-hour and 4-hour postprandial glucose (PPG [meal test]) was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period. Meal test: The subjects were given a carbohydrate-rich standardised liquid meal immediately after bolus (faster aspart or NovoRapid®) infusion in the morning of the meal test. The subjects were to consume the meal as quickly as possible (within 12 minutes) and blood samples were drawn after 30 minutes, 1, 2, 3 and 4 hours from the start of the meal.
Time Frame: Week 0, week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L
  30-min (Baseline): number analyzed (Participants) | 236 | 234
  30-min (Baseline) | 10.54 (3.33) | 10.30 (2.96)
  1-hour (Baseline): number analyzed (Participants) | 235 | 235
  1-hour (Baseline) | 12.18 (3.96) | 11.96 (3.81)
  2-hour (Baseline): number analyzed (Participants) | 236 | 235
  2-hour (Baseline) | 13.17 (4.77) | 13.04 (4.35)
  3-hour (Baseline): number analyzed (Participants) | 235 | 233
  3-hour (Baseline) | 11.38 (4.65) | 11.48 (4.28)
  4-hour (Baseline): number analyzed (Participants) | 233 | 231
  4-hour (Baseline) | 9.07 (4.31) | 9.18 (3.83)
  30-min (Change from baseline): number analyzed (Participants) | 229 | 226
  30-min (Change from baseline) | -0.50 (4.05) | 0.42 (3.75)
  1-hour (Change from baseline): number analyzed (Participants) | 228 | 229
  1-hour (Change from baseline) | -0.85 (4.65) | 0.36 (4.58)
  2-hour (Change from baseline): number analyzed (Participants) | 230 | 227
  2-hour (Change from baseline) | -0.80 (5.33) | 0.42 (5.01)
  3-hour (Change from baseline): number analyzed (Participants) | 228 | 226
  3-hour (Change from baseline) | -0.33 (5.12) | 0.20 (4.75)
  4-hour (Change from baseline): number analyzed (Participants) | 225 | 223
  4-hour (Change from baseline) | 0.00 (4.76) | 0.21 (4.10)

9. Secondary Outcome: Change From Baseline in 30-min, 2-hour, 3-hour and 4-hour PPG Increment (Meal Test)
Description: Change from baseline (week 0) in 30-min, 2-hour, 3-hour and 4-hour PPG increment (meal test) was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period. Meal test: The subjects were given a carbohydrate-rich standardised liquid meal immediately after bolus (faster aspart or NovoRapid®) infusion in the morning of the meal test. The subjects were to consume the meal as quickly as possible (within 12 minutes) and PPG was evaluated after 30 minutes, 1, 2, 3 and 4 hours from the start of the meal.
Time Frame: Week 0, week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L
  30-min (Baseline): number analyzed (Participants) | 236 | 234
  30-min (Baseline) | 3.02 (2.16) | 2.95 (2.03)
  2-hour (Baseline): number analyzed (Participants) | 236 | 235
  2-hour (Baseline) | 5.65 (4.12) | 5.70 (3.66)
  3-hour (Baseline): number analyzed (Participants) | 235 | 233
  3-hour (Baseline) | 3.85 (4.32) | 4.13 (3.72)
  4-hour (Baseline): number analyzed (Participants) | 233 | 231
  4-hour (Baseline) | 1.57 (4.23) | 1.83 (3.52)
  30-min (Change from baseline): number analyzed (Participants) | 229 | 224
  30-min (Change from baseline) | -0.53 (2.47) | 0.11 (2.25)
  2-hour (Change from baseline): number analyzed (Participants) | 230 | 225
  2-hour (Change from baseline) | -0.82 (4.39) | 0.09 (4.13)
  3-hour (Change from baseline): number analyzed (Participants) | 228 | 224
  3-hour (Change from baseline) | -0.35 (4.53) | -0.14 (4.07)
  4-hour (Change from baseline): number analyzed (Participants) | 225 | 221
  4-hour (Change from baseline) | 0.01 (4.50) | -0.11 (3.76)

10. Secondary Outcome: Change From Baseline in Mean of the 7-7-9 Point Self-measured Plasma Glucose (SMPG) Profile
Description: Change from baseline (week 0) in mean of the 7-7-9 point SMPG profile was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period. 7-7-9 point SMPG was measured at the following mentioned time points: 1) Before breakfast, 2) 60 mins after the start of Breakfast, 3) Before lunch, 4) 60 mins after the start of lunch, 5) Before main evening meal, 6) 60 mins after the start of main evening meal, 7) At bedtime, 8) At 4 AM, 9) Before breakfast.
Time Frame: Week 0, week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L
  Baseline: number analyzed (Participants) | 208 | 209
  Baseline | 9.24 (1.71) | 9.10 (1.40)
  Change from baseline: number analyzed (Participants) | 196 | 196
  Change from baseline | 0.19 (1.91) | 0.10 (1.58)

11. Secondary Outcome: Change From Baseline of the 7-7-9 Point SMPG Profile: PPG (Mean, Breakfast, Lunch and Main Evening Meal)
Description: Change from baseline (week 0) in PPG (breakfast, lunch, main evening meal and mean over all meals) of the 7-7-9 point SMPG profile was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L
  Breakfast (baseline): number analyzed (Participants) | 188 | 189
  Breakfast (baseline) | 10.82 (2.99) | 10.28 (3.07)
  Lunch (baseline): number analyzed (Participants) | 191 | 197
  Lunch (baseline) | 9.65 (3.05) | 9.62 (2.68)
  Main evening meal (baseline): number analyzed (Participants) | 194 | 194
  Main evening meal (baseline) | 9.79 (3.01) | 9.34 (3.06)
  Mean over all meals (baseline): number analyzed (Participants) | 168 | 171
  Mean over all meals (baseline) | 10.07 (2.09) | 9.74 (1.99)
  Breakfast (Change from baseline): number analyzed (Participants) | 177 | 176
  Breakfast (Change from baseline) | -0.33 (3.61) | 0.23 (3.79)
  Lunch (Change from baseline): number analyzed (Participants) | 177 | 181
  Lunch (Change from baseline) | 0.27 (3.75) | 0.05 (3.57)
  Main evening meal (Change from baseline): number analyzed (Participants) | 174 | 175
  Main evening meal (Change from baseline) | -0.35 (3.81) | 0.58 (3.61)
  Mean over all meals (Change from baseline): number analyzed (Participants) | 147 | 152
  Mean over all meals (Change from baseline) | 0.06 (2.33) | 0.13 (2.21)

12. Secondary Outcome: Change From Baseline of the 7-7-9 Point SMPG Profile: PPG Increment (Mean, Breakfast, Lunch and Main Evening Meal)
Description: Change from baseline (week 0) in PPG increment (breakfast, lunch, main evening meal and mean over all meals) of the 7-7-9 point SMPG profile was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L
  Breakfast (baseline): number analyzed (Participants) | 182 | 184
  Breakfast (baseline) | 2.62 (3.16) | 1.93 (3.28)
  Lunch (baseline): number analyzed (Participants) | 186 | 189
  Lunch (baseline) | 1.80 (2.77) | 1.77 (2.47)
  Main evening meal (baseline): number analyzed (Participants) | 186 | 191
  Main evening meal (baseline) | 1.04 (3.07) | 0.52 (2.69)
  Mean over all meals (baseline): number analyzed (Participants) | 156 | 164
  Mean over all meals (baseline) | 1.93 (1.94) | 1.48 (1.86)
  Breakfast (Change from baseline): number analyzed (Participants) | 167 | 167
  Breakfast (Change from baseline) | -0.75 (3.90) | 0.03 (3.67)
  Lunch (Change from baseline): number analyzed (Participants) | 171 | 171
  Lunch (Change from baseline) | -0.43 (3.25) | -0.27 (3.13)
  Main evening meal (Change from baseline): number analyzed (Participants) | 163 | 171
  Main evening meal (Change from baseline) | -0.47 (3.51) | 0.35 (3.79)
  Mean over all meals (Change from baseline): number analyzed (Participants) | 131 | 139
  Mean over all meals (Change from baseline) | -0.53 (1.99) | 0.12 (1.92)

13. Secondary Outcome: Change From Baseline of the 7-7-9 Point SMPG Profile: Pre-prandial Plasma Glucose (PG) (Mean, Pre-breakfast, Pre-lunch, Pre-main Evening Meal)
Description: Change from baseline (week 0) in pre-prandial PG (pre-breakfast, pre-lunch, pre-main evening meal and mean over all meals) of the 7-7-9 point SMPG profile was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L
  Pre-breakfast (baseline): number analyzed (Participants) | 204 | 206
  Pre-breakfast (baseline) | 8.40 (2.50) | 8.31 (2.32)
  Pre-lunch (baseline): number analyzed (Participants) | 207 | 207
  Pre-lunch (baseline) | 8.28 (2.85) | 8.21 (2.32)
  Pre-main evening meal (baseline): number analyzed (Participants) | 203 | 208
  Pre-main evening meal (baseline) | 8.68 (2.76) | 8.87 (2.62)
  Pre-mean over all meals (baseline): number analyzed (Participants) | 199 | 205
  Pre-mean over all meals (baseline) | 8.39 (1.73) | 8.45 (1.54)
  Pre-breakfast (Change from baseline): number analyzed (Participants) | 192 | 192
  Pre-breakfast (Change from baseline) | 0.36 (3.33) | 0.26 (3.05)
  Pre-lunch (Change from baseline): number analyzed (Participants) | 195 | 193
  Pre-lunch (Change from baseline) | 0.39 (3.54) | 0.21 (3.12)
  Pre-main evening meal (Change from baseline): number analyzed (Participants) | 189 | 194
  Pre-main evening meal (Change from baseline) | 0.15 (3.72) | 0.13 (3.18)
  Pre-mean over all meals (Change from baseline): number analyzed (Participants) | 185 | 189
  Pre-mean over all meals (Change from baseline) | 0.39 (2.00) | 0.21 (1.84)

14. Secondary Outcome: Change From Baseline of the 7-7-9 Point SMPG Profile: Fluctuation in 7-7-9 Point Profile
Description: Fluctuation in 7-point SMPG profile was the average absolute difference from the mean of the SMPG profile. Reported results are fluctuation in the 7-7-9 point SMPG profile at baseline (week 0) and after 16 weeks of randomisation (i.e., week 16). The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Median (Full Range); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L
  Baseline: number analyzed (Participants) | 208 | 209
  Baseline | 2.14 [0.4 to 4.9] | 2.05 [0.9 to 4.0]
  Last in-trial value: number analyzed (Participants) | 212 | 214
  Last in-trial value | 2.06 [0.9 to 5.2] | 2.06 [0.7 to 3.8]

15. Secondary Outcome: Change From Baseline of the 7-7-9 Point SMPG Profile: in Nocturnal SMPG Measurements
Description: Change from baseline (week 0) in nocturnal SMPG measurements was assessed by considering the differences between PG values available at bedtime, at 4 AM and the before breakfast value the following day: (4 AM PG value minus at bedtime PG value), (before breakfast PG value minus at bedtime PG value) and (before breakfast PG value minus 4 AM PG value). Change from baseline in nocturnal increments in SMPG measurements of the 7-7-9 point SMPG profile was evaluated after 16 weeks of randomisation and presented during three different time intervals as follows: 1) 04:00 to breakfast, 2) bedtime to 04:00, and 3) bedtime to breakfast. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L
  04:00 to breakfast (Baseline): number analyzed (Participants) | 176 | 181
  04:00 to breakfast (Baseline) | -1.29 (3.61) | -1.06 (3.35)
  Bedtime to 04:00 (Baseline): number analyzed (Participants) | 167 | 174
  Bedtime to 04:00 (Baseline) | -0.97 (5.16) | -0.56 (3.84)
  Bedtime to breakfast (Baseline): number analyzed (Participants) | 193 | 195
  Bedtime to breakfast (Baseline) | -1.73 (4.81) | -1.56 (3.83)
  04:00 to breakfast (Change from baseline): number analyzed (Participants) | 152 | 165
  04:00 to breakfast (Change from baseline) | -0.50 (4.83) | -0.08 (4.45)
  Bedtime to 04:00 (Change from baseline): number analyzed (Participants) | 144 | 155
  Bedtime to 04:00 (Change from baseline) | 0.81 (6.59) | 0.18 (5.14)
  Bedtime to breakfast (Change from baseline): number analyzed (Participants) | 182 | 179
  Bedtime to breakfast (Change from baseline) | 0.13 (6.67) | -0.20 (5.84)

16. Secondary Outcome: Percentage of Subjects Reaching Overall PPG (1 Hour) ≤7.8 mmol/L [140 mg/dL]
Description: Percentage of subjects reaching overall PPG (1 hour) ≤7.8 mmol/L [140 mg/dL] was evaluated after 16 weeks of randomisation. Subjects without a postprandial glucose measurement at week 16 were considered not to have achieved HbA1c target at week 16. The results are based on the in-trial period.
Time Frame: Week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Number; unit: % of subjects
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
% of subjects | 8.1 | 7.6

17. Secondary Outcome: Percentage of Subjects Reaching Overall PPG (1 Hour) ≤7.8 mmol/L [140 mg/dL] Without Severe Hypoglycaemia
Description: Percentage of subjects reaching overall PPG (1 hour) ≤7.8 mmol/L [140 mg/dL] without treatment emergent severe hypoglycaemia was evaluated after 16 weeks of randomisation. Subjects without a postprandial glucose measurement at week 16 were considered not to have achieved HbA1c target at week 16. Severe hypoglycaemia: An episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. Plasma glucose (PG) concentrations may not be available during an event, but neurological recovery following the return of PG to normal was considered sufficient evidence that the event was induced by a low PG concentration. The results are based on the in-trial period.
Time Frame: Week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Number; unit: % of subjects
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
% of subjects | 7.6 | 6.8

18. Secondary Outcome: Change From Baseline in Lipids-lipoproteins Profile (Total Cholesterol, High Density Lipoproteins, Low Density Lipoproteins)
Description: Reported results are lipids-lipoproteins (total cholesterol, high density lipoproteins, low density lipoproteins) values at baseline (week 0) and after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Median (Full Range); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L
  Total cholesterol (Baseline) | 4.48 [2.6 to 8.1] | 4.68 [2.9 to 8.0]
  High density lipoproteins (Baseline) | 1.70 [0.8 to 3.3] | 1.71 [0.8 to 3.8]
  Low density lipoproteins (Baseline) | 2.46 [1.1 to 6.4] | 2.63 [1.2 to 6.6]
  Total cholesterol (Last in-trial value) | 4.61 [2.8 to 7.2] | 4.57 [2.4 to 8.2]
  High density lipoproteins (Last in-trial value) | 1.74 [0.9 to 3.1] | 1.74 [0.7 to 3.6]
  Low density lipoproteins (Last in-trial value) | 2.56 [1.0 to 5.2] | 2.59 [1.1 to 6.4]

19. Secondary Outcome: Insulin Dose in Units/Day: Total Basal
Description: Total basal insulin dose (Units/day) was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period: the observation period from date of first dose of randomised trial products (faster aspart and NovoRapid®) to no later than 7 days after the day of last dose of randomised trial products.
Time Frame: Week 16
Population: The safety analysis set included all subjects receiving at least one dose of the investigational medicinal product (IMP, faster aspart) or its comparator (NovoRapid®/NovoLog®). Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: Unit (U)
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Unit (U) | 23.82 (12.82) | 23.87 (11.38)

20. Secondary Outcome: Insulin Dose in Units/Day: Total Bolus
Description: Total bolus insulin dose (Units/day) was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 16
Population: The safety analysis set included all subjects receiving at least one dose of the IMP or its comparator. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: U
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
U | 25.91 (17.46) | 25.27 (15.33)

21. Secondary Outcome: Insulin Dose in Units/Day: Total Daily Insulin Dose
Description: Total insulin dose (Units/day) was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: U
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
U | 49.72 (27.08) | 49.12 (23.75)

22. Secondary Outcome: Insulin Dose in Units/Day: Individual Meal Insulin Dose
Description: No data was collected for individual meal insulin dose.
Time Frame: Week 16
Population: No subjects were analysed, as no data was collected for individual meal insulin dose.
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Insulin Dose in Units/kg/Day: Total Basal
Description: Total basal insulin dose (Units/kg/day) was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: U/Kg
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
U/Kg | 0.30 (0.12) | 0.30 (0.11)

24. Secondary Outcome: Insulin Dose in Units/kg/Day: Total Bolus
Description: Total bolus insulin dose (Units/kg/day) was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: U/Kg
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
U/Kg | 0.33 (0.17) | 0.31 (0.16)

25. Secondary Outcome: Insulin Dose in Units/kg/Day: Total Daily Insulin Dose
Description: Total insulin dose (Units/kg/day) was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: U/Kg
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
U/Kg | 0.63 (0.24) | 0.61 (0.23)

26. Secondary Outcome: Insulin Dose in Units/kg/Day: Individual Meal Insulin Dose
Description: No data was collected for individual meal insulin dose.
Time Frame: Week 16
Population: No subjects were analysed, as no data was collected for individual meal insulin dose.
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Insulin Delivery Pump Parameter: Insulin Carbohydrate Ratio
Description: Insulin carbohydrate ratio was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Gram (g)/U
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Gram (g)/U | 9.13 (3.20) | 9.74 (6.77)

28. Secondary Outcome: Insulin Delivery Pump Parameter: Glucose Sensitivity Factor
Description: Glucose sensitivity factor was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mmol/L/U
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L/U | 2.65 (1.14) | 2.60 (0.98)

29. Secondary Outcome: Insulin Delivery Pump Parameter: Active Insulin Time
Description: Active insulin time was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Hour (h)
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Hour (h) | 3.6 (0.7) | 3.6 (0.7)

30. Secondary Outcome: Change From Baseline in Mean IG Increment (0-30 Min, 0-1 Hour and 0-2 Hours After Start of Meal) (Mean, Breakfast, Lunch and Main Evening Meal)
Description: Change from baseline (week 0) in mean interstitial glucose (IG) increment (0-30 minutes (min), 0-1 hour (h) and 0-2 h after start of meal) (breakfast, lunch, main evening meal and mean across all meals) was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L
  Breakfast 0-30 min (Baseline): number analyzed (Participants) | 229 | 230
  Breakfast 0-30 min (Baseline) | 0.23 (0.61) | 0.21 (0.60)
  Lunch 0-30 min (Baseline): number analyzed (Participants) | 230 | 231
  Lunch 0-30 min (Baseline) | 0.02 (0.54) | 0.03 (0.60)
  Main evening meal 0-30 min (Baseline): number analyzed (Participants) | 231 | 231
  Main evening meal 0-30 min (Baseline) | 0.15 (0.52) | 0.09 (0.57)
  Mean across all meals 0-30 min (Baseline): number analyzed (Participants) | 228 | 230
  Mean across all meals 0-30 min (Baseline) | 0.13 (0.37) | 0.11 (0.39)
  Breakfast 0-1 h (Baseline): number analyzed (Participants) | 229 | 230
  Breakfast 0-1 h (Baseline) | 0.78 (0.97) | 0.73 (0.94)
  Lunch 0-1 h (Baseline): number analyzed (Participants) | 230 | 231
  Lunch 0-1 h (Baseline) | 0.42 (0.77) | 0.44 (0.84)
  Main evening meal 0-1 h (Baseline): number analyzed (Participants) | 231 | 231
  Main evening meal 0-1 h (Baseline) | 0.39 (0.75) | 0.32 (0.82)
  Mean across all meals 0-1 h (Baseline): number analyzed (Participants) | 228 | 230
  Mean across all meals 0-1 h (Baseline) | 0.52 (0.57) | 0.50 (0.60)
  Breakfast 0-2 h (Baseline): number analyzed (Participants) | 229 | 230
  Breakfast 0-2 h (Baseline) | 1.32 (1.52) | 1.27 (1.46)
  Lunch 0-2 h (Baseline): number analyzed (Participants) | 230 | 231
  Lunch 0-2 h (Baseline) | 0.99 (1.19) | 0.92 (1.07)
  Main evening meal 0-2 h (Baseline): number analyzed (Participants) | 231 | 231
  Main evening meal 0-2 h (Baseline) | 0.54 (1.15) | 0.50 (1.19)
  Mean across all meals 0-2 h (Baseline): number analyzed (Participants) | 228 | 230
  Mean across all meals 0-2 h (Baseline) | 0.93 (0.94) | 0.89 (0.84)
  Breakfast 0-30 min (Change from baseline): number analyzed (Participants) | 225 | 221
  Breakfast 0-30 min (Change from baseline) | -0.03 (0.80) | 0.08 (0.67)
  Lunch 0-30 min (Change from baseline): number analyzed (Participants) | 226 | 223
  Lunch 0-30 min (Change from baseline) | 0.05 (0.61) | 0.10 (0.68)
  Main evening meal 0-30 min (Change from baseline): number analyzed (Participants) | 227 | 223
  Main evening meal 0-30 min (Change from baseline) | -0.07 (0.73) | -0.01 (0.70)
  Mean across all meals 0-30min:Change from baseline: number analyzed (Participants) | 224 | 221
  Mean across all meals 0-30min:Change from baseline | -0.01 (0.46) | 0.06 (0.46)
  Breakfast 0-1 h (Change from baseline): number analyzed (Participants) | 225 | 221
  Breakfast 0-1 h (Change from baseline) | -0.13 (1.13) | 0.14 (0.99)
  Lunch 0-1 h (Change from baseline): number analyzed (Participants) | 226 | 223
  Lunch 0-1 h (Change from baseline) | -0.02 (0.88) | 0.15 (0.99)
  Main evening meal 0-1 h (Change from baseline): number analyzed (Participants) | 227 | 223
  Main evening meal 0-1 h (Change from baseline) | -0.16 (0.95) | 0.04 (0.97)
  Mean across all meals 0-1 h (Change from baseline): number analyzed (Participants) | 224 | 221
  Mean across all meals 0-1 h (Change from baseline) | -0.10 (0.61) | 0.11 (0.66)
  Breakfast 0-2 h (Change from baseline): number analyzed (Participants) | 225 | 221
  Breakfast 0-2 h (Change from baseline) | -0.28 (1.60) | 0.16 (1.45)
  Lunch 0-2 h (Change from baseline): number analyzed (Participants) | 226 | 223
  Lunch 0-2 h (Change from baseline) | -0.24 (1.32) | 0.22 (1.37)
  Main evening meal 0-2 h (Change from baseline): number analyzed (Participants) | 227 | 223
  Main evening meal 0-2 h (Change from baseline) | -0.29 (1.29) | -0.03 (1.27)
  Mean across all meals 0-2 h (Change from baseline): number analyzed (Participants) | 224 | 221
  Mean across all meals 0-2 h (Change from baseline) | -0.25 (0.81) | 0.12 (0.86)

31. Secondary Outcome: Change From Baseline in Mean Time to the IG Peak After Start of Meal (Mean, Breakfast, Lunch and Main Evening Meal)
Description: Change from baseline (week 0) in mean time to the IG peak after start of meal (breakfast, lunch, main evening meal and mean across all meals) was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Minutes
  Breakfast (Baseline): number analyzed (Participants) | 229 | 231
  Breakfast (Baseline) | 88.95 (25.66) | 97.29 (32.32)
  Lunch (Baseline): number analyzed (Participants) | 230 | 231
  Lunch (Baseline) | 109.47 (31.78) | 106.94 (29.67)
  Main evening meal (Baseline): number analyzed (Participants) | 231 | 232
  Main evening meal (Baseline) | 110.11 (32.35) | 106.91 (29.61)
  Mean across all meals (Baseline): number analyzed (Participants) | 231 | 232
  Mean across all meals (Baseline) | 103.24 (18.50) | 103.99 (19.21)
  Breakfast (Change from baseline): number analyzed (Participants) | 225 | 222
  Breakfast (Change from baseline) | 0.25 (33.69) | -4.03 (35.49)
  Lunch (Change from baseline): number analyzed (Participants) | 226 | 223
  Lunch (Change from baseline) | -2.00 (38.63) | 1.64 (38.02)
  Main evening meal (Change from baseline): number analyzed (Participants) | 227 | 223
  Main evening meal (Change from baseline) | -2.04 (40.51) | -1.43 (38.94)
  Mean across all meals (Change from baseline): number analyzed (Participants) | 227 | 223
  Mean across all meals (Change from baseline) | -1.30 (22.01) | -1.00 (21.90)

32. Secondary Outcome: Change From Baseline in Mean IG Peak After Start of Meal (Mean, Breakfast, Lunch and Main Evening Meal)
Description: Change from baseline (week 0) in mean IG peak after start of meal (breakfast, lunch, main evening meal and mean across all meals) was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L
  Breakfast (Baseline): number analyzed (Participants) | 229 | 231
  Breakfast (Baseline) | 12.43 (1.97) | 12.25 (2.09)
  Lunch (Baseline): number analyzed (Participants) | 230 | 231
  Lunch (Baseline) | 12.42 (2.07) | 12.56 (1.84)
  Main evening meal (Baseline): number analyzed (Participants) | 231 | 232
  Main evening meal (Baseline) | 12.65 (2.10) | 12.70 (2.06)
  Mean across all meals (Baseline): number analyzed (Participants) | 231 | 232
  Mean across all meals (Baseline) | 12.49 (1.67) | 12.51 (1.60)
  Breakfast (Change from baseline): number analyzed (Participants) | 225 | 222
  Breakfast (Change from baseline) | 0.10 (2.24) | 0.11 (2.11)
  Lunch (Change from baseline): number analyzed (Participants) | 226 | 223
  Lunch (Change from baseline) | 0.10 (2.19) | 0.19 (1.92)
  Main evening meal (Change from baseline): number analyzed (Participants) | 227 | 223
  Main evening meal (Change from baseline) | 0.22 (2.09) | -0.13 (2.14)
  Mean across all meals (Change from baseline): number analyzed (Participants) | 227 | 223
  Mean across all meals (Change from baseline) | 0.16 (1.63) | 0.03 (1.59)

33. Secondary Outcome: Percentage of Time Spent With IG ≤2.5, 3.0, 3.5, 3.9 mmol/L [45, 54, 63, 70 mg/dL]) and IG >10.0, 12.0, 13.9 mmol/L [180, 216, 250 mg/dL])
Description: Percentage of time spent with IG ≤2.5, 3.0, 3.5, 3.9 mmol/L [45, 54, 63, 70 mg/dL]) and IG >10.0, 12.0, 13.9 mmol/L [180, 216, 250 mg/dL]) was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: % of time
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
% of time
  IG ≤2.5 mmol/L (45 mg/dL): number analyzed (Participants) | 234 | 231
  IG ≤2.5 mmol/L (45 mg/dL) | 1.11 (1.29) | 1.03 (1.38)
  IG ≤3.0 mmol/L (54 mg/dL): number analyzed (Participants) | 234 | 231
  IG ≤3.0 mmol/L (54 mg/dL) | 2.15 (1.98) | 2.19 (2.25)
  IG ≤3.5 mmol/L (63 mg/dL): number analyzed (Participants) | 234 | 231
  IG ≤3.5 mmol/L (63 mg/dL) | 3.75 (2.85) | 3.93 (3.37)
  IG ≤3.9 mmol/L (70.2 mg/dL): number analyzed (Participants) | 234 | 231
  IG ≤3.9 mmol/L (70.2 mg/dL) | 5.46 (3.68) | 5.76 (4.25)
  IG >10.0 mmol/L (180 mg/dL): number analyzed (Participants) | 234 | 231
  IG >10.0 mmol/L (180 mg/dL) | 41.57 (13.09) | 39.24 (11.86)
  IG >12.0 mmol/L (216 mg/dL): number analyzed (Participants) | 234 | 231
  IG >12.0 mmol/L (216 mg/dL) | 26.34 (11.66) | 24.23 (10.75)
  IG >13.9 mmol/L (250 mg/dL): number analyzed (Participants) | 234 | 231
  IG >13.9 mmol/L (250 mg/dL) | 15.87 (9.42) | 14.23 (8.49)

34. Secondary Outcome: Incidence of Episodes With IG ≤2.5, 3.0, 3.5, 3.9 mmol/L [45, 54, 63, 70 mg/dL]) and IG >10.0, 12.0, 13.9 mmol/L [180, 216, 250 mg/dL])
Description: Incidence of episodes with IG ≤2.5, 3.0, 3.5, 3.9 mmol/L [45, 54, 63, 70 mg/dL]) and IG >10.0, 12.0, 13.9 mmol/L [180, 216, 250 mg/dL]) was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Number; unit: Number of Events
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of Events
  IG ≤2.5 mmol/L (45 mg/dL): number analyzed (Participants) | 208 | 205
  IG ≤2.5 mmol/L (45 mg/dL) | 1570 | 1532
  IG ≤3.0 mmol/L (54 mg/dL): number analyzed (Participants) | 226 | 222
  IG ≤3.0 mmol/L (54 mg/dL) | 2848 | 2920
  IG ≤3.5 mmol/L (63 mg/dL): number analyzed (Participants) | 232 | 227
  IG ≤3.5 mmol/L (63 mg/dL) | 4584 | 4742
  IG ≤3.9 mmol/L (70 mg/dL): number analyzed (Participants) | 234 | 229
  IG ≤3.9 mmol/L (70 mg/dL) | 6371 | 6576
  IG >10.0 mmol/L (180 mg/dL): number analyzed (Participants) | 234 | 231
  IG >10.0 mmol/L (180 mg/dL) | 35194 | 33176
  IG >12.0 mmol/L (216 mg/dL): number analyzed (Participants) | 234 | 231
  IG >12.0 mmol/L (216 mg/dL) | 23070 | 21276
  IG >13.9 mmol/L (250 mg/dL): number analyzed (Participants) | 234 | 231
  IG >13.9 mmol/L (250 mg/dL) | 14352 | 12866

35. Secondary Outcome: Change From Baseline in Mean of the IG Profile
Description: Change from baseline (week 0) in mean of the IG profile was evaluated after 16 weeks of randomisation. The mean of an IG profile is defined as the time integral of the profile over the profile's length, divided by the profile's length. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L
  Baseline | 9.38 (1.18) | 9.39 (1.20)
  Change from baseline: number analyzed (Participants) | 234 | 231
  Change from baseline | 0.28 (1.27) | 0.04 (1.18)

36. Secondary Outcome: Percentage of Time Spent Within IG Target Range 4.0-7.8 mmol/L (71-140 mg/dL) and 4.0-10 mmol/L (71-180 mg/dL)
Description: Percentage of time spent within IG target range 4.0-7.8 mmol/L (71-140 mg/dL) and 4.0-10 mmol/L (71-180 mg/dL) was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: % of time
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
% of time
  IG 4.0-7.8 mmol/L (71-140 mg/dL): number analyzed (Participants) | 234 | 231
  IG 4.0-7.8 mmol/L (71-140 mg/dL) | 31.49 (9.97) | 33.11 (8.76)
  IG 4.0-10.0 mmol/L (71-180 mg/dL): number analyzed (Participants) | 234 | 231
  IG 4.0-10.0 mmol/L (71-180 mg/dL) | 52.40 (11.87) | 54.40 (10.70)

37. Secondary Outcome: Variation in the IG Profile
Description: Variation in IG profile was the average absolute difference from the mean of the IG profile. Variation in the IG profile was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Median (Full Range); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L | 3.09 [1.6 to 5.6] | 3.04 [1.6 to 5.1]

38. Secondary Outcome: Area Under the Curve (AUC3.9-IG) for IG ≤3.9 mmol/L [70 mg/dL]
Description: Area under the curve (AUC3.9-IG) for IG ≤3.9 mmol/L [70 mg/dL] was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L | 3.19 (0.22) | 3.21 (0.20)

39. Secondary Outcome: Change From Baseline in AUCIG,0-15min
Description: Change from baseline (week 0) in area under the curve for interstitial glucose (AUCIG),0-15 minutes during meal test was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L
  Baseline: number analyzed (Participants) | 221 | 228
  Baseline | 7.55 (2.63) | 7.37 (2.20)
  Change from baseline: number analyzed (Participants) | 203 | 198
  Change from baseline | 0.16 (3.06) | 0.21 (2.96)

40. Secondary Outcome: Change From Baseline in AUCIG,0-30min
Description: Change from baseline (week 0) in AUCIG,0-30 minutes during meal test was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L
  Baseline: number analyzed (Participants) | 221 | 228
  Baseline | 7.98 (2.65) | 7.86 (2.25)
  Change from baseline: number analyzed (Participants) | 205 | 198
  Change from baseline | 0.12 (3.12) | 0.22 (3.02)

41. Secondary Outcome: Change From Baseline in AUCIG,0-1h
Description: Change from baseline (week 0) in AUCIG,0-1 hour during meal test was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L
  Baseline: number analyzed (Participants) | 221 | 228
  Baseline | 9.47 (2.76) | 9.35 (2.38)
  Change from baseline: number analyzed (Participants) | 207 | 200
  Change from baseline | -0.07 (3.33) | 0.32 (3.26)

42. Secondary Outcome: Change From Baseline in AUCIG,0-2h
Description: Change from baseline (week 0) in AUCIG,0-2 hours during meal test was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L
  Baseline: number analyzed (Participants) | 225 | 228
  Baseline | 11.27 (3.10) | 11.18 (2.82)
  Change from baseline: number analyzed (Participants) | 211 | 206
  Change from baseline | -0.38 (3.76) | 0.37 (3.90)

43. Secondary Outcome: Change From Baseline in AUCIG,0-4h
Description: Change from baseline (week 0) in AUCIG,0-24hours during meal test was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L
  Baseline: number analyzed (Participants) | 226 | 229
  Baseline | 11.31 (3.33) | 11.40 (3.03)
  Change from baseline: number analyzed (Participants) | 215 | 210
  Change from baseline | -0.32 (4.07) | 0.29 (4.10)

44. Secondary Outcome: Change From Baseline in Time to the IG Peak After Start of Meal
Description: Change from baseline (week 0) in time to the IG peak after start of meal-test meal was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: Minute
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Minute
  Baseline: number analyzed (Participants) | 226 | 229
  Baseline | 111.2 (45.3) | 117.0 (43.0)
  Change from baseline: number analyzed (Participants) | 215 | 210
  Change from baseline | 1.2 (50.5) | -1.4 (51.6)

45. Secondary Outcome: Change From Baseline in IG Peak After Start of Meal
Description: Change from baseline (week 0) in IG peak after start of meal-test meal was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Week 0, week 16
Population: The FAS included all randomised subjects. Number analyzed = Number of subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L
  Baseline: number analyzed (Participants) | 226 | 229
  Baseline | 14.71 (3.94) | 14.69 (3.65)
  Change from baseline: number analyzed (Participants) | 215 | 210
  Change from baseline | -0.57 (4.69) | 0.36 (4.78)

46. Secondary Outcome: Number of Treatment Emergent Adverse Events (AEs)
Description: Treatment emergent adverse events (TEAEs) were recorded from week 0 to week 16. A TEAE was defined as an event that has an onset date on or after the first day of exposure to randomised treatment (in week 0), and no later than seven days after the last day of randomised treatment (i.e., maximum week 16 + 7 days). The results are based on the on-treatment period.
Time Frame: Weeks 0-16
Population: as for outcome 20
Measure: Number; unit: Number of adverse events
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of adverse events | 440 | 412

47. Secondary Outcome: Number of Treatment Emergent Infusion Site Reactions
Description: Number of treatment emergent infusion site reactions were recorded from week 0 to week 16. The results are based on the on-treatment period.
Time Frame: Weeks 0-16
Population: as for outcome 20
Measure: Number; unit: Number of infusion site reaction events
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of infusion site reaction events | 44 | 32

48. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to the American Diabetes Association (ADA) and Novo Nordisk (NN) Definition: Overall
Description: ADA classification of hypo:
  1. Severe: Requiring assistance of another person to actively administer carbohydrate/glucagon/take other corrective actions. PG levels may not be available during an event, but neurological recovery following return of PG to normal is considered sufficient evidence that event was induced by a low PG level.
  2. Documented symptomatic: PG ≤3.9 mmol/L with symptoms.
  3. Asymptomatic: PG ≤3.9 mmol/L without symptoms.
  4. Probable symptomatic: No measurement with symptoms.
  5. Pseudo: PG >3.9 mmol/L with symptoms.
  6. Unclassifiable.
  NN classification of hypo:
  1. BG confirmed: PG <3.1 mmol/L with/without symptoms.
  2. Severe or BG confirmed symptomatic: Severe as per ADA and BG confirmed by PG <3.1 mmol/L with symptoms.
  3. Severe or BG confirmed: Severe as per ADA and BG confirmed by PG <3.1 mmol/L with/without symptoms.
  4. Unclassifiable.
  Not able to self treat-unclassifiable: Not able to self treat but not classifiable as severe hypo.
Time Frame: Weeks 0-16
Population: The safety analysis set included all subjects receiving at least one dose of the IMP or its comparator. Number analyzed = Number of subjects contributed to the analysis. The results are based on the on-treatment period.
Measure: Number; unit: Number of hypoglycaemic episodes
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of hypoglycaemic episodes
  ADA: Severe | 21 | 7
  ADA: Documented symptomatic | 8372 | 8904
  ADA: Asymptomatic | 2530 | 2273
  ADA: Probable symptomatic | 88 | 32
  ADA: Pseudo | 56 | 159
  ADA: Unclassifiable | 1 | 0
  NN: BG confirmed | 3258 | 3240
  NN: Severe or BG confirmed symptomatic | 2751 | 2779
  NN: Severe or BG confirmed | 3279 | 3247
  NN: Unclassifiable | 7789 | 8128
  Not able to selftreat - unclassifiable | 0 | 0

49. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to the American Diabetes Association and Novo Nordisk Definition: Daytime Hypoglycaemic Episodes (06:00-00:00 - Inclusive)
Description: Number of treatment emergent day time hypoglycaemic episodes according to the ADA and NN definitions were evaluated between 06:00 and 00:00 (both included). The results are based on the on-treatment period.
Time Frame: Weeks 0-16
Population: as for outcome 20
Measure: Number; unit: Number of hypoglycaemic episodes
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of hypoglycaemic episodes
  ADA: Severe | 12 | 5
  ADA: Documented symptomatic | 7508 | 7889
  ADA: Asymptomatic | 2321 | 2071
  ADA: Probable symptomatic | 70 | 26
  ADA: Pseudo | 52 | 144
  ADA: Unclassifiable | 0 | 0
  NN: BG confirmed | 2799 | 2769
  NN: Severe or BG confirmed symptomatic | 2335 | 2359
  NN: Severe or BG confirmed | 2811 | 2774
  NN: Unclassifiable | 7152 | 7361
  Not able to selftreat - unclassifiable | 0 | 0

50. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to the American Diabetes Association and Novo Nordisk Definition: Nocturnal Hypoglycaemic Episodes (00:01-05:59 - Inclusive)
Description: Number of treatment emergent nocturnal hypoglycaemic episodes according to the ADA and NN definitions were evaluated between 00:01 and 05:59 (both included). The results are based on the on-treatment period.
Time Frame: Weeks 0-16
Population: as for outcome 20
Measure: Number; unit: Number of hypoglycaemic episodes
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of hypoglycaemic episodes
  ADA: Severe | 9 | 2
  ADA: Documented symptomatic | 864 | 1015
  ADA: Asymptomatic | 209 | 202
  ADA: Probable symptomatic | 18 | 6
  ADA: Pseudo | 4 | 15
  ADA: Unclassifiable | 1 | 0
  NN: BG confirmed | 459 | 471
  NN: Severe or BG confirmed symptomatic | 416 | 420
  NN: Severe or BG confirmed | 468 | 473
  NN: Unclassifiable | 637 | 767
  Not able to selftreat - unclassifiable | 0 | 0

51. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to the American Diabetes Association and Novo Nordisk Definition: Hypoglycaemic Episodes During First 1 Hour After Start of the Meal
Description: Number of treatment emergent hypoglycaemic episodes according to the ADA and NN definitions were evaluated during the first 1 hour after start of the meal. The results are based on the on-treatment period.
Time Frame: Weeks 0-16
Population: as for outcome 20
Measure: Number; unit: Number of hypoglycaemic episodes
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of hypoglycaemic episodes
  ADA: Severe | 0 | 0
  ADA: Documented symptomatic | 224 | 190
  ADA: Asymptomatic | 31 | 33
  ADA: Probable symptomatic | 1 | 3
  ADA: Pseudo | 0 | 5
  ADA: Unclassifiable | 0 | 0
  NN: BG confirmed | 92 | 51
  NN: Severe or BG confirmed symptomatic | 81 | 48
  NN: Severe or BG confirmed | 92 | 51
  NN: Unclassifiable | 164 | 180
  Not able to selftreat - unclassifiable | 0 | 0

52. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to the American Diabetes Association and NN Definition: Hypoglycaemic Episodes During First 2 Hours After Start of the Meal
Description: Number of treatment emergent hypoglycaemic episodes according to the ADA and NN definitions were evaluated during the first 2 hours after start of the meal. The results are based on the on-treatment period.
Time Frame: Weeks 0-16
Population: as for outcome 20
Measure: Number; unit: Number of hypoglycaemic episodes
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of hypoglycaemic episodes
  ADA: Severe | 0 | 0
  ADA: Documented symptomatic | 1258 | 1077
  ADA: Asymptomatic | 176 | 175
  ADA: Probable symptomatic | 9 | 6
  ADA: Pseudo | 7 | 34
  ADA: Unclassifiable | 0 | 0
  NN: BG confirmed | 482 | 413
  NN: Severe or BG confirmed symptomatic | 441 | 372
  NN: Severe or BG confirmed | 482 | 413
  NN: Unclassifiable | 968 | 879
  Not able to selftreat - unclassifiable | 0 | 0

53. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to the American Diabetes Association and NN Definition: Hypoglycaemic Episodes During First 4 Hours After Start of the Meal
Description: Number of treatment emergent hypoglycaemic episodes according to the ADA and NN definitions were evaluated during the first 4 hours after start of the meal. The results are based on the on-treatment period.
Time Frame: Weeks 0-16
Population: as for outcome 20
Measure: Number; unit: Number of hypoglycaemic episodes
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of hypoglycaemic episodes
  ADA: Severe | 5 | 2
  ADA: Documented symptomatic | 3767 | 3907
  ADA: Asymptomatic | 750 | 677
  ADA: Probable symptomatic | 43 | 17
  ADA: Pseudo | 29 | 98
  ADA: Unclassifiable | 0 | 0
  NN: BG confirmed | 1403 | 1399
  NN: Severe or BG confirmed symptomatic | 1246 | 1259
  NN: Severe or BG confirmed | 1408 | 1401
  NN: Unclassifiable | 3186 | 3300
  Not able to selftreat - unclassifiable | 0 | 0

54. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to the American Diabetes Association and NN Definition: Hypoglycaemic Episodes Occurring Between 2 to 4 Hours After Start of the Meal
Description: Number of treatment emergent hypoglycaemic episodes according to the ADA and NN definitions were evaluated between 2 to 4 hours after start of the meal. The results are based on the on-treatment period.
Time Frame: Weeks 0-16
Population: as for outcome 20
Measure: Number; unit: Number of hypoglycaemic episodes
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of hypoglycaemic episodes
  ADA: Severe | 5 | 2
  ADA: Documented symptomatic | 2509 | 2830
  ADA: Asymptomatic | 574 | 502
  ADA: Probable symptomatic | 34 | 11
  ADA: Pseudo | 22 | 64
  ADA: Unclassifiable | 0 | 0
  NN: BG confirmed | 921 | 986
  NN: Severe or BG confirmed symptomatic | 805 | 887
  NN: Severe or BG confirmed | 926 | 988
  NN: Unclassifiable | 2218 | 2421
  Not able to selftreat - unclassifiable | 0 | 0

55. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to the American Diabetes Association and NN Definition: Hypoglycaemic Episodes Occurring Between 1 Hour to 2 Hours After Start of the Meal
Description: Number of treatment emergent hypoglycaemic episodes according to the ADA and NN definitions were evaluated between 1 hour to 2 hours after start of the meal. The results are based on the on-treatment period.
Time Frame: Weeks 0-16
Population: as for outcome 20
Measure: Number; unit: Number of hypoglycaemic episodes
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of hypoglycaemic episodes
  ADA: Severe | 0 | 0
  ADA: Documented symptomatic | 1034 | 887
  ADA: Asymptomatic | 145 | 142
  ADA: Probable symptomatic | 8 | 3
  ADA: Pseudo | 7 | 29
  ADA: Unclassifiable | 0 | 0
  NN: BG confirmed | 390 | 362
  NN: Severe or BG confirmed symptomatic | 360 | 324
  NN: Severe or BG confirmed | 390 | 362
  NN: Unclassifiable | 804 | 699
  Not able to selftreat - unclassifiable | 0 | 0

56. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to the American Diabetes Association and Novo Nordisk Definition: Hypoglycaemic Episodes Occurring Between 2 to 3 Hours After Start of the Meal
Description: Number of treatment emergent hypoglycaemic episodes according to the ADA and NN definitions were evaluated between 2 to 3 hours after start of the meal. The results are based on the on-treatment period.
Time Frame: Weeks 0-16
Population: as for outcome 20
Measure: Number; unit: Number of hypoglycaemic episodes
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of hypoglycaemic episodes
  ADA: Severe | 2 | 1
  ADA: Documented symptomatic | 1327 | 1518
  ADA: Asymptomatic | 277 | 241
  ADA: Probable symptomatic | 19 | 7
  ADA: Pseudo | 13 | 38
  ADA: Unclassifiable | 0 | 0
  NN: BG confirmed | 491 | 555
  NN: Severe or BG confirmed symptomatic | 429 | 508
  NN: Severe or BG confirmed | 493 | 556
  NN: Unclassifiable | 1145 | 1249
  Not able to selftreat - unclassifiable | 0 | 0

57. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to the American Diabetes Association and Novo Nordisk Definition: Hypoglycaemic Episodes Occurring Between 3 to 4 Hours After Start of the Meal
Description: Number of treatment emergent hypoglycaemic episodes according to the ADA and NN definitions were evaluated between 3 to 4 hours after start of the meal. The results are based on the on-treatment period.
Time Frame: Weeks 0-16
Population: as for outcome 20
Measure: Number; unit: Number of hypoglycaemic episodes
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of hypoglycaemic episodes
  ADA: Severe | 3 | 1
  ADA: Documented symptomatic | 1182 | 1312
  ADA: Asymptomatic | 297 | 261
  ADA: Probable symptomatic | 15 | 4
  ADA: Pseudo | 9 | 26
  ADA: Unclassifiable | 0 | 0
  NN: BG confirmed | 430 | 431
  NN: Severe or BG confirmed symptomatic | 376 | 379
  NN: Severe or BG confirmed | 433 | 432
  NN: Unclassifiable | 1073 | 1172
  Not able to selftreat - unclassifiable | 0 | 0

58. Secondary Outcome: Number of Unexplained Episodes of Hyperglycaemia (Confirmed by SMPG)
Description: Unexplained hyperglycaemia was defined as a confirmed PG value ≥16.7 mmol/L (300 mg/dL) and was unexplained (i.e. no apparent medical, dietary, insulin dosage or pump failure reason). The results are based on the on-treatment period.
Time Frame: Weeks 0-16
Population: as for outcome 20
Measure: Number; unit: Number of hypoglycaemic episodes
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of hypoglycaemic episodes | 1185 | 1058

59. Secondary Outcome: Change From Baseline in Physical Examination: Respiratory System
Description: Reported results are respiratory system-examination findings at baseline (week 0) and after 16 weeks of randomisation. The findings are presented as: 1) Normal. 2) Abnormal (not clinically significant [NCS]). 3) Abnormal (clinically significant [CS]). The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Number; unit: Number of subjects
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of subjects
  Normal, baseline | 234 | 235
  Abnormal (NCS), baseline | 1 | 1
  Abnormal (CS), baseline | 1 | 0
  Normal, last on-treatment value | 235 | 234
  Abnormal (NCS), last on-treatment value | 0 | 2
  Abnormal (CS), last on-treatment value | 1 | 0

60. Secondary Outcome: Change From Baseline in Physical Examination: Cardiovascular System
Description: Reported results are cardiovascular system-examination findings at baseline (week 0) and after 16 weeks of randomisation. The findings are presented as: 1) Normal. 2) Abnormal (not clinically significant [NCS]). 3) Abnormal (clinically significant [CS]). The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Number; unit: Number of subjects
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of subjects
  Normal, baseline | 233 | 229
  Abnormal (NCS), baseline | 1 | 7
  Abnormal (CS), baseline | 2 | 0
  Normal, last on-treatment value | 231 | 228
  Abnormal (NCS), last on-treatment value | 4 | 7
  Abnormal (CS), last on-treatment value | 1 | 1

61. Secondary Outcome: Change From Baseline in Physical Examination: Central and Peripheral Nervous System
Description: Reported results are central and peripheral nervous system-examination findings at baseline (week 0) and after 16 weeks of randomisation. The findings are presented as: 1) Normal. 2) Abnormal (not clinically significant [NCS]). 3) Abnormal (clinically significant [CS]). The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Number; unit: Number of subjects
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of subjects
  Normal, baseline | 210 | 215
  Abnormal (NCS), baseline | 22 | 18
  Abnormal (CS), baseline | 4 | 3
  Normal, last on-treatment value | 209 | 216
  Abnormal (NCS), last on-treatment value | 23 | 17
  Abnormal (CS), last on-treatment value | 4 | 3

62. Secondary Outcome: Change From Baseline in Physical Examination: Gastrointestinal System, Including the Mouth
Description: Reported results are gastrointestinal system-examination findings at baseline (week 0) and after 16 weeks of randomisation. The findings are presented as: 1) Normal. 2) Abnormal (not clinically significant [NCS]). 3) Abnormal (clinically significant [CS]). The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Number; unit: Number of subjects
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of subjects
  Normal, baseline | 231 | 231
  Abnormal (NCS), baseline | 3 | 5
  Abnormal (CS), baseline | 2 | 0
  Normal, last on-treatment value | 231 | 231
  Abnormal (NCS), last on-treatment value | 4 | 3
  Abnormal (CS), last on-treatment value | 1 | 2

63. Secondary Outcome: Change From Baseline in Physical Examination: Musculoskeletal System
Description: Reported results are musculoskeletal system-examination findings at baseline (week 0) and after 16 weeks of randomisation. The findings are presented as: 1) Normal. 2) Abnormal (not clinically significant [NCS]). 3) Abnormal (clinically significant [CS]). The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Number; unit: Number of subjects
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of subjects
  Normal, baseline | 222 | 227
  Abnormal (NCS), baseline | 13 | 9
  Abnormal (CS), baseline | 1 | 0
  Normal, last on-treatment value | 223 | 228
  Abnormal (NCS), last on-treatment value | 12 | 8
  Abnormal (CS), last on-treatment value | 1 | 0

64. Secondary Outcome: Change From Baseline in Physical Examination: Skin
Description: Reported results are skin-examination findings at baseline (week 0) and after 16 weeks of randomisation. The findings are presented as: 1) Normal. 2) Abnormal (not clinically significant [NCS]). 3) Abnormal (clinically significant [CS]). The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Number; unit: Number of subjects
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of subjects
  Normal, baseline | 212 | 211
  Abnormal (NCS), baseline | 18 | 22
  Abnormal (CS), baseline | 6 | 3
  Normal, last on-treatment value | 204 | 203
  Abnormal (NCS), last on-treatment value | 21 | 29
  Abnormal (CS), last on-treatment value | 11 | 4

65. Secondary Outcome: Change From Baseline in Physical Examination: Head, Ears, Eyes, Nose, Throat and Neck
Description: Reported results are head, ears, eyes, nose, throat and neck-examination findings at baseline (week 0) and after 16 weeks of randomisation. The findings are presented as: 1) Normal. 2) Abnormal (not clinically significant [NCS]). 3) Abnormal (clinically significant [CS]). The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Number; unit: Number of subjects
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of subjects
  Normal, baseline | 219 | 221
  Abnormal (NCS), baseline | 15 | 14
  Abnormal (CS), baseline | 2 | 1
  Normal, last on-treatment value | 217 | 218
  Abnormal (NCS), last on-treatment value | 15 | 16
  Abnormal (CS), last on-treatment value | 4 | 2

66. Secondary Outcome: Change From Baseline in Vital Sign: Blood Pressure
Description: Change from baseline (week 0) in blood pressure (both systolic and diastolic) was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmHg
  Systolic blood pressure (baseline) | 123.6 (14.7) | 122.0 (14.3)
  Diastolic blood pressure (baseline) | 74.8 (9.4) | 74.6 (8.7)
  Systolic blood pressure (change from baseline) | -0.8 (12.3) | -0.7 (11.5)
  Diastolic blood pressure (change from baseline) | -0.7 (8.4) | -0.4 (7.7)

67. Secondary Outcome: Change From Baseline in Vital Sign: Pulse
Description: Change from baseline (week 0) in pulse was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Beats/minute
  Baseline | 73.7 (11.0) | 74.5 (11.1)
  Change from baseline | -0.5 (9.0) | -0.8 (9.6)

68. Secondary Outcome: Change From Screening in Electrocardiogram (ECG)
Description: Reported results are ECG findings at screening (week -6) and after 16 weeks of randomisation. The findings are presented as: 1) Normal. 2) Abnormal (not clinically significant [NCS]). 3) Abnormal (clinically significant [CS]). The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Number; unit: Number of subjects
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of subjects
  Normal, screening | 178 | 181
  Abnormal (NCS), screening | 58 | 54
  Abnormal (CS), screening | 0 | 1
  Normal, last on-treatment value: number analyzed (Participants) | 232 | 230
  Normal, last on-treatment value | 188 | 180
  Abnormal (NCS), last on-treatment value: number analyzed (Participants) | 232 | 230
  Abnormal (NCS), last on-treatment value | 44 | 48
  Abnormal (CS), last on-treatment value: number analyzed (Participants) | 232 | 230
  Abnormal (CS), last on-treatment value | 0 | 2

69. Secondary Outcome: Change From Screening in Fundus Photography/Fundoscopy
Description: Reported results are fundus photography/fundoscopy (for both left and right eye) findings at screening (week -6) and after 16 weeks of randomisation. The findings are presented as: 1) Normal. 2) AAbnormal (not clinically significant [NCS]). 3) Abnormal (clinically significant [CS]). The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Number; unit: Number of subjects
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of subjects
  Left eye (Normal), screening | 135 | 136
  Left eye (Abnormal [NCS]), screening | 94 | 94
  Left eye (Abnormal [CS]), screening | 7 | 6
  Right eye (Normal), screening | 132 | 132
  Right eye (Abnormal [NCS]), screening | 98 | 98
  Right eye (Abnormal [CS]), screening | 6 | 6
  Left eye (Normal), last on-treatment value: number analyzed (Participants) | 217 | 208
  Left eye (Normal), last on-treatment value | 130 | 119
  Left eye (Abnormal [NCS]), last on-treatment value: number analyzed (Participants) | 217 | 208
  Left eye (Abnormal [NCS]), last on-treatment value | 77 | 82
  Left eye (Abnormal [CS] last on-treatment value: number analyzed (Participants) | 217 | 208
  Left eye (Abnormal [CS] last on-treatment value | 10 | 7
  Right eye (Normal), last on-treatment value: number analyzed (Participants) | 217 | 208
  Right eye (Normal), last on-treatment value | 127 | 114
  Right eye (Abnormal-NCS), last on-treatment value: number analyzed (Participants) | 217 | 208
  Right eye (Abnormal-NCS), last on-treatment value | 80 | 87
  Right eye (Abnormal [CS]), last on-treatment value: number analyzed (Participants) | 217 | 208
  Right eye (Abnormal [CS]), last on-treatment value | 10 | 7

70. Secondary Outcome: Change From Baseline in Haematology: Haemoglobin
Description: Change from baseline (week 0) in haemoglobin was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L
  Baseline | 8.62 (0.82) | 8.62 (0.80)
  Change from baseline | -0.01 (0.48) | -0.06 (0.40)

71. Secondary Outcome: Change From Baseline in Haematology: Haematocrit
Description: Change from baseline (week 0) in haematocrit was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: % of haematocrit
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
% of haematocrit
  Baseline | 42.23 (3.98) | 42.37 (3.77)
  Change from baseline | 0.09 (2.47) | -0.30 (2.01)

72. Secondary Outcome: Change From Baseline in Haematology: Erythrocytes
Description: Change from baseline (week 0) in erythrocytes was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: 10^12/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
10^12/L
  Baseline | 4.66 (0.45) | 4.72 (0.42)
  Change from baseline | 0.01 (0.27) | -0.03 (0.22)

73. Secondary Outcome: Change From Baseline in Haematology: Thrombocytes
Description: Change from baseline (week 0) in thrombocytes was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
10^9/L
  Baseline | 246.4 (58.9) | 243.6 (55.3)
  Change from baseline | 2.2 (33.5) | 0.2 (35.8)

74. Secondary Outcome: Change From Baseline in Haematology: Leucocytes
Description: Change from baseline (week 0) in leucocytes was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
10^9/L
  Baseline | 6.41 (1.78) | 6.32 (1.70)
  Change from baseline | -0.09 (1.49) | -0.03 (1.22)

75. Secondary Outcome: Change From Baseline in Biochemistry: Total Protein
Description: Change from baseline (week 0) in total protein was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
g/dL
  Baseline | 6.73 (0.44) | 6.74 (0.47)
  Change from baseline | 0.03 (0.36) | -0.05 (0.40)

76. Secondary Outcome: Change From Baseline in Biochemistry: Creatinine
Description: Change from baseline (week 0) in creatinine was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
umol/L
  Baseline | 73.8 (12.3) | 74.5 (13.3)
  Change from baseline | 0.9 (7.9) | -0.1 (8.2)

77. Secondary Outcome: Change From Baseline in Biochemistry: Alanine Aminotransferase (ALT)
Description: Change from baseline (week 0) in ALT was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
U/L
  Baseline | 20.0 (11.6) | 19.1 (11.5)
  Change from baseline | 0.1 (13.8) | 0 (9.4)

78. Secondary Outcome: Change From Baseline in Biochemistry: Aspartate Aminotransferase (AST)
Description: Change from baseline (week 0) in AST was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
U/L
  Baseline | 22.2 (9.1) | 20.6 (7.8)
  Change from baseline | -0.1 (18.6) | -0.4 (8.7)

79. Secondary Outcome: Change From Baseline in Biochemistry: Alkaline Phosphatase (ALP)
Description: Change from baseline (week 0) in ALP was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
U/L
  Baseline | 68.8 (20.8) | 69.7 (23.9)
  Change from baseline | 1.2 (9.6) | 0.8 (10.0)

80. Secondary Outcome: Change From Baseline in Biochemistry: Sodium
Description: Change from baseline (week 0) in sodium was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L
  Baseline | 140.3 (2.7) | 140.3 (2.7)
  Change from baseline | -0.2 (2.9) | -0.2 (2.5)

81. Secondary Outcome: Change From Baseline in Biochemistry: Potassium
Description: Change from baseline (week 0) in potassium was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mmol/L
  Baseline | 4.34 (0.42) | 4.30 (0.39)
  Change from baseline | -0.02 (0.42) | -0.01 (0.41)

82. Secondary Outcome: Change From Baseline in Biochemistry: Albumin
Description: Change from baseline (week 0) in albumin was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
g/dL
  Baseline | 4.32 (0.27) | 4.31 (0.28)
  Change from baseline | -0.01 (0.22) | -0.05 (0.26)

83. Secondary Outcome: Change From Baseline in Biochemistry: Total Bilirubin
Description: Change from baseline (week 0) in bilirubin was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
umol/L
  Baseline | 8.2 (5.1) | 8.8 (6.4)
  Change from baseline | -0.3 (3.8) | -1.0 (3.7)

84. Secondary Outcome: Change From Baseline in Urinalysis: Albumin/Creatine Ratio
Description: Change from baseline (week 0) in albumin/creatine ratio was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mg/mmol
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
mg/mmol
  Baseline | 2.67 (13.88) | 2.00 (7.60)
  Change from baseline | 0.01 (4.76) | -0.04 (3.11)

85. Secondary Outcome: Change From Baseline in Urinalysis: Erythrocytes
Description: Reported results are urine erythrocytes-test findings at baseline (week 0) and after 16 weeks of randomisation. The findings are presented as: a) Negative, b) Trace, c) 1+, d) 2+ and e) 3+. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Number; unit: Number of subjects
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of subjects
  Negative (baseline) | 217 | 215
  Trace (baseline) | 8 | 10
  1+ (baseline) | 5 | 5
  2+ (baseline) | 5 | 1
  3+ (baseline) | 1 | 5
  Negative (last on-treatment value) | 217 | 215
  Trace (last on-treatment value) | 6 | 10
  1+ (last on-treatment value) | 3 | 3
  2+ (last on-treatment value) | 2 | 4
  3+ (last on-treatment value) | 8 | 4

86. Secondary Outcome: Change From Baseline in Urinalysis: Protein
Description: Reported results are urine protein-test findings at baseline (week 0) and after 16 weeks of randomisation. The findings are presented as: a) Negative, b) Trace, c) 1+, d) 2+ e) 3+ and f) 4+. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Number; unit: Number of subjects
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of subjects
  Negative (baseline) | 193 | 195
  Trace (baseline) | 31 | 27
  1+ (baseline) | 8 | 10
  2+ (baseline) | 4 | 4
  3+ (baseline) | 0 | 0
  4+ (baseline) | 0 | 0
  Negative (last on-treatment value) | 196 | 196
  Trace (last on-treatment value) | 27 | 27
  1+ (last on-treatment value) | 10 | 9
  2+ (last on-treatment value) | 2 | 4
  3+ (last on-treatment value) | 1 | 0
  4+ (last on-treatment value) | 0 | 0

87. Secondary Outcome: Change From Baseline in Urinalysis: Ketones
Description: Reported results are urine ketone-test findings at baseline (week 0) and after 16 weeks of randomisation. The findings are presented as: a) Negative, b) Trace, c) 1+, d) 2+ e) 3+ and f) 4+. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Number; unit: Number of subjects
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of subjects
  Negative (baseline) | 192 | 205
  Trace (baseline) | 31 | 23
  1+ (baseline) | 11 | 8
  2+ (baseline) | 2 | 0
  3+ (baseline) | 0 | 0
  4+ (baseline) | 0 | 0
  Negative (last on-treatment value) | 194 | 203
  Trace (last on-treatment value) | 25 | 27
  1+ (last on-treatment value) | 15 | 5
  2+ (last on-treatment value) | 2 | 1
  3+ (last on-treatment value) | 0 | 0
  4+ (last on-treatment value) | 0 | 0

88. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline (week 0) in body weight was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Kg
  Baseline | 76.86 (15.20) | 78.21 (14.47)
  Change from baseline | 0.34 (1.90) | 0.80 (2.14)

89. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: Change from baseline (week 0) in BMI was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
kg/m^2
  Baseline | 26.16 (4.06) | 26.51 (3.89)
  Change from baseline | 0.12 (0.65) | 0.28 (0.74)

90. Secondary Outcome: Number of Change-of-infusion-sets Per Week
Description: Number of change-of-infusion-sets per week was evaluated from week 0 to week 16. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: Week 0-16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Number of infusion-sets
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of infusion-sets | 2.55 (0.43) | 2.49 (0.47)

91. Secondary Outcome: Number of Subjects With at Least One Non-routine Change-of-infusion-sets Categorised by Reasons for Change-of-infusion-sets
Description: Number of subjects with at least one non-routine change-of-infusion-sets categorised by reasons for change-of-infusion-sets was evaluated from week 0 to week 16. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
  Reasons for change-of-infusion-sets are categorised as follows:
  Category-1: A perceived occlusion by the subject Category-2: Any problems related to the infusion set Category-3: Any technical issues with the pump Category-4: Changes in the insulin solution in the infusion set or reservoir Category-5: High BG with no other explanation which made the subject change the infusion set Category-6: Infusion site reaction Category-7: Missing
Time Frame: Week 0-16
Population: as for outcome 20
Measure: Number; unit: Number of subjects
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 236 | 236
Number of subjects
  Category-1 | 50 | 50
  Category-2 | 108 | 75
  Category-3 | 23 | 17
  Category-4 | 3 | 8
  Category-5 | 66 | 60
  Category-6 | 16 | 8
  Category-7 | 3 | 1

ADVERSE EVENTS:
Time Frame: Week 0 to Week 16 + 7 days. All reported AEs are treatment emergent (i.e., TEAE).
Description: Results are based on the safety analysis set, which included all subjects receiving at least one dose of the IMP or its comparator.
Arm/Group | Faster Aspart | NovoRapid
All-Cause Mortality (participants affected / at risk) | 0/236 | 0/236
Serious Adverse Events (participants affected / at risk) | 5/236 | 8/236
Other Adverse Events (participants affected / at risk) | 84/236 | 72/236
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Faster Aspart (N=236) | NovoRapid (N=236)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Device breakage (Product Issues) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 (1) | 1 (1)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain management (Surgical and medical procedures) | 0 (0) | 1 (1)
Retinal aneurysm (Eye disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Faster Aspart (N=236) | NovoRapid (N=236)
Gastroenteritis (Infections and infestations) | 12 (12) | 6 (6)
Infusion site reaction (General disorders) | 16 (26) | 7 (10)
Upper respiratory tract infection (Infections and infestations) | 17 (18) | 12 (12)
Viral upper respiratory tract infection (Infections and infestations) | 48 (60) | 50 (64)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT02825251/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT02825251/SAP_001.pdf